CLINICAL TRIAL: NCT02649387
Title: Minimal Residual Disease Eradication With Ibrutinib Therapy (MERIT) in Patients With Chronic Lymphocytic Leukemia After Frontline Therapy
Brief Title: Ibrutinib in Treating Minimal Residual Disease in Patients With Chronic Lymphocytic Leukemia After Front-Line Therapy
Acronym: MERIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1481; NCI-2015-02153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-004991 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Results first posted 2025-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Treatment repeats every 4 weeks* for up to 36 courses in the absence of disease progression or unacceptable toxicity.
  Note: *The last course may last up to 56 days to accommodate the study drug discontinuation visit.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well ibrutinib works in treating patients with chronic lymphocytic leukemia who responded to initial treatment used to reduce a cancer (front-line therapy) but have residual disease. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the rate of minimal residual disease (MRD)-negative responses (in both blood and bone marrow) at any time during treatment with ibrutinib maintenance.

SECONDARY OBJECTIVES:

I. Median time to achieve MRD- (negative) status (in blood and in bone marrow) after initiation of ibrutinib maintenance treatment.

II. Toxicity profile of ibrutinib as maintenance therapy after frontline induction.

III. Durability of the MRD- state (determined from the time of first documentation of MRD- until the first documentation of MRD+ (positive) (or last date shown to be MRD- for a censor).

IV. Determine the number of patients who improve their remission category (i.e., upgrade clinical response achieved after the induction such as from partial response [PR] to complete response [CR]) after initiating the maintenance therapy.

V. Time to requirement of next therapy for patients who achieve confirmed MRD- vs. those who remain MRD+ disease at 48 weeks (end of 12 cycles).

VI. Progression free survival (as determined by the International Workshop on Chronic Lymphocytic Leukemia [IWCLL] criteria) among patients who achieve confirmed MRD- vs. those who remain MRD+ disease at 48 weeks (end of 12 cycles).

TERTIARY OBJECTIVES:

I. To conduct correlative studies for further understanding of the mechanism of antitumor activity of ibrutinib in eradication of the MRD.

II. Determine the impact of ibrutinib on depression and anxiety symptoms to better understand toxicity profile of ibrutinib maintenance.

III. Determine impact of social support or lack thereof on mood symptoms in chronic lymphocytic leukemia (CLL) patients receiving maintenance treatment.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 4 weeks* for up to 36 courses in the absence of disease progression or unacceptable toxicity.

Note: *The last course may last up to 56 days to accommodate the study drug discontinuation visit.

After completion of study treatment, patients are followed up every 3-6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements including willing to provide blood, baseline bone marrow aspirate, and control deoxyribonucleic acid (DNA) samples for correlative research purposes
* Diagnosis of B-cell chronic lymphocytic leukemia (B-CLL), confirmed by flow cytometry and as per the criteria outlined by the IWCLL/Hallek December 2008
* Prior frontline therapy for B-CLL must have been discontinued >= 56 days but =< 365 days prior to registration; NOTE: Patients on supportive care therapy due to use of specific induction regimen such as antibiotics may continue on those treatments at the discretion of the treating physician
* Patient must have completed a frontline induction therapy (minimum of 2 treatment cycles); NOTE: Standard therapies/therapeutic agents are defined as those listed in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of CLL; also, patients who received induction regimen as part of a clinical trial and is not necessarily mentioned in the NCCN guidelines, will also be eligible as long as the patient has completed at least 2 treatment cycles of induction regimen, achieved a clinical response (PR or CR) and is able to meet all other criteria for the study; however, patients who have previously received ibrutinib or have been randomized to ibrutinib containing arms in a clinical trial will not be eligible for this study
* Patients must have a sustained clinical response (PR, nodular PR [nPR], complete clinical response [CCR], CR with incomplete marrow recovery [CRi], CR) with documented residual disease (>= 1 CLL cell per 10,000 leukocytes or >= 0.01% MRD) either in the blood, bone marrow or a lymph node >= 3.5 cm by any available techniques
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 at registration
* Absolute neutrophil count >= 1000/mm^3
* Platelet count >= 30,000/mm^3
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 mg/dL or direct bilirubin =< 1.0 mg/dL for patients with Gilbert's syndrome
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3.5 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Since this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown, any of the following will deem the subject ineligible for the study:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy =< 28 days prior to registration on this study; NOTE: Patients on low dose prednisone (=< 10 mg) for treatment of conditions other than CLL are eligible
* Patients who have received more than 1 prior therapy; NOTE: Prior therapy is defined as any single agent or combination regimen that is included as treatment for symptomatic CLL; treatment(s) given prior to the symptomatic phase of the disease (preventive strategy) will not be considered as prior induction therapy; for the purpose of a particular therapy/regimen to be counted towards the number of prior treatments a patient must have received at least 2 cycles of the induction regimen e.g., a patient who change their treatment regimen after only 1 cycle (due to toxicity or any other reason) will not be considered to have "2" prior therapies
* Patients who have progressive disease or relapse (as defined by the IWCLL criteria) at or any time before registration on this study
* Patients with history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off therapy for that disease for > 3 years)
* Patients who are already MRD- (both in the blood and the bone marrow) after frontline therapy and have lymph nodes < 3.5 cm
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 modulators (cytochrome P450, family 3, subfamily A [CYP3A] inhibitor and/or CYP3A inducers)
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Major surgery =< 4 weeks prior to registration
* Patients who have active infectious hepatitis
* Patients with other diseases that in the opinion of the treating physician pose a higher risk for treatment with ibrutinib therapy including active human immunodeficiency virus (HIV) infection and bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2026-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher Chanan-Khan, M.D., Principal Investigator — Mayo Clinic; Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ibrutinib): Patients receive ibrutinib PO QD on days 1-28. Treatment repeats every 4 weeks* for up to 36 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Confirmed MRD-negative Response
Description: This outcome is summarized by the proportion of patients achieving MRD negative status. A confirmed MRD-negative response is defined as an achievement of MRD-negative status in both the blood and the bone marrow on two consecutive evaluations at least 3 months apart.
Time Frame: 3 years
Measure: Number; unit: proportion of patients
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 35
proportion of patients | 0

2. Secondary Outcome: Duration of MRD-negative Response
Description: Defined as the time from the earliest date that the patient was noted as having MRD-negative response in both the blood and bone marrow until the first notation of MRD positive disease in the blood or the bone marrow.
Time Frame: 5 years
Population: No patients achieved MRD status, thus no patients are evaluable for this outcome measure.
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Improvement in Clinical Response
Description: Assessed using International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Adverse Events
Description: Will be graded according to the Grading Scale for Hematologic Adverse Events in CLL Studies. The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Time Frame: Up to 30 days after the last day of study drug treatment
Reporting Status: Not Posted

5. Secondary Outcome: Progression-free Survival
Description: Defined as the time from the 48-week MRD evaluation until the time of disease progression per the IWCLL criteria or death due to any cause
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Time to MRD-negative Response
Description: Defined as the time from the date of registration to the earliest date that the patient was noted as having MRD-negative response in both the blood and bone marrow
Time Frame: 5 years
Population: No patients achieved MRD status, thus no patients are evaluable for this outcome measure.
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Requirement of Next Therapy
Description: Defined as the time from the 48-week MRD evaluation until the time of initiation of subsequent treatment for progressive CLL
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 3 years and mortality was followed for 8 years
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 16/35
Other Adverse Events (participants affected / at risk) | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=35)
Anemia (Blood and lymphatic system disorders) | 14 (59)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 6 (10)
Skin infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (3)
Wound infection (Infections and infestations) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5)
Lymphocyte count increased (Investigations) | 9 (135)
Neutrophil count decreased (Investigations) | 10 (33)
Platelet count decreased (Investigations) | 24 (326)
White blood cell decreased (Investigations) | 7 (14)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Headache (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 10 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT02649387/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02649387/ICF_001.pdf